CLINICAL TRIAL: NCT03545997
Title: Impact of Blocked Cysteinyl Leukotriene Pathway on Endothelial Function in Patients With Obstructive Sleep Apnea Syndrome: Multicenter Randomized Placebo Controlled Crossover Trial
Brief Title: Montelukast for Patients With Obstructive Sleep Apnea Syndrome
Acronym: MONTSAS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Act For Chronic Diseases (Other); Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 38RC17.107
Record Dates: First submitted 2018-05-16; First posted 2018-06-06 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Montelukast; leukotriene pathway; endothelial function; flux-mediated dilation
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — montelukast

STUDY DESIGN:
Intervention Model Description: It's a prospective, randomized, comparative vs placebo, double blind, multicenter, national study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Montelukast will be crushed and coated in a capsule, Mannitol is into a capsule too.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Montelukast (Experimental): Drug :Montelukast, capsule, 10mg, one per day in the evening, one hour before or 2 hours post meal, length of treatment 3 months
  Interventions: Drug: Montelukast 10mg; Drug: Placebo
- Placebo (Placebo Comparator): Drug: Mannitol, capsule, 350mg, one per day in the evening, one hour before or 2 hours post meal, length of treatment 3 months
  Interventions: Drug: Montelukast 10mg; Drug: Placebo

INTERVENTIONS:
Drug: Montelukast 10mg — The capsules will be presented in box of 95 capsules packaged in unit blister
Drug: Placebo — Mannitol 350mg The capsules will be presented in box of 95 capsules packaged in unit blister

SUMMARY:
This study compares the effect of Montelukast vs Placebo on Flow Mediated Dilatation of the Brachial Artery (FMD) in patients with obstructive sleep apnea syndrome.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea Syndrome (OSAS) induces low-grade systemic and vascular inflammation, including activation of the leukotriene pathway.

In apneic patients, the urinary excretion of LTE4, a systemic marker of CysLT pathway activation, is increased in relation to the severity of OSAS and it's an independent predictor of cardiovascular risk event occurring at 10 years.

Montelukast is a CysLT1 receptor antagonist. By blocking CysLT1 receptors, montelukast prevents vasoconstriction, proliferation and migration of smooth muscle cells, adhesion molecule expression, and leukocyte recruitment induced by CysLTs.Montelukast may improve endothelial function and reduce vascular remodeling in apneic patients.

A pharmacological blockade of CysLT pathway would be an interesting therapeutic strategy to limit the cardiovascular consequences of OSAS.

ELIGIBILITY:
Inclusion Criteria:

* With mild to moderate obstructive sleep apnea syndrome (apnea / hypopnea index> 15 and <30 events per hour)
* Little symptomatic (Epworth sleepiness score <10)
* Polysomnography within 3 months prior to inclusion
* With a history of myocardial infarction or stroke
* Affiliation to Social Security or beneficiary of such a scheme
* Signed consent

Exclusion Criteria:

* OSAS support by PPC
* Cancer
* Chronic inflammatory disease
* Asthma previously treated with Montelukast
* Chronic infectious disease
* Epworth sleepiness scale ≥10
* Contraindication to Montelukast: Hypersensitivity to the active substance or to the excipients
* Contraindications to trinitrin: hypersensitivity to nitrates, state of shock, severe hypotension, association with sildenafil, obstructive cardiomyopathy, inferior right sided myocardial infarction with right ventricular extension, acute, except in case of signs left ventricular failure, intracranial hypertension, breastfeeding
* Treatment with phenobarbital, phenytoin, rifampicin: risk of montelukast metabolism increase and thus decrease of its effectiveness
* Persons referred in Articles L1121-5 to L1121-8 of the CSP (pregnant woman, parturient, nursing mothers, person deprived of liberty by judicial or administrative decision, person subject to a measure of legal protection, can not be included in clinical trials)
* Subject in exclusion period of another study
* Subject can not be contacted in case of emergency

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Change in FMD of the brachial artery between the beginning and end of each treatment period (Montelukast and placebo), expressed as absolute value (FMD unit is %) and measured in a standardized manner. | before and after 3 months treatment

SECONDARY OUTCOMES:
Concentrations of urinary LTE4 at the beginning and end of each treatment period | before and after 3 months the two periods of treatment
24h ambulatory blood pressure (systolic and diastolic) measurement | before and after 3 months of the two periods of treatment, and 15 days after the last period
Polysomnography at inclusion and at the end of each treatment period | inclusion and at the end of the two periods of treatment
Plasma concentration of Montelukast measured by HPLC-MS at the end of the Montelukast treatment period | at the end of Montelukast treatment period
Collection of adverse events | from inclusion to 15 days after the last period of treatment
Comparison of Cardiovascular Events occurence (myocardial infarction, Stroke, Cardiovascular Death) between the two periods | from inclusion to 15 days after the last period of treatment
Concentrations of plasma CRPus at baseline and at the beginning and end of each treatment period | before and after 3 months the two periods of treatment

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - University Hospital, Bron
  - Métropole Savoie Hospital, Chambéry
  - University Hospital, Clermont-Ferrand
  - University Hospital Grenoble, Grenoble
  - University Hospital, Grenoble
  - Annecy Genevois Hospital, Metz-Tessy
  - University Hospital, Pierre-Bénite
  - University Hospital, Saint-Etienne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ingelsson E, Yin L, Back M. Nationwide cohort study of the leukotriene receptor antagonist montelukast and incident or recurrent cardiovascular disease. J Allergy Clin Immunol. 2012 Mar;129(3):702-707.e2. doi: 10.1016/j.jaci.2011.11.052. Epub 2012 Jan 12. PMID 22244598
- [Background] Goldbart AD, Greenberg-Dotan S, Tal A. Montelukast for children with obstructive sleep apnea: a double-blind, placebo-controlled study. Pediatrics. 2012 Sep;130(3):e575-80. doi: 10.1542/peds.2012-0310. Epub 2012 Aug 6. PMID 22869829
- [Background] Cereza G, Garcia Dolade N, Laporte JR. Nightmares induced by montelukast in children and adults. Eur Respir J. 2012 Dec;40(6):1574-5. doi: 10.1183/09031936.00092812. No abstract available. PMID 23204025
- [Background] Marchand MS, Jonville-Bera AP, Autret-Leca E; Association francaise des centres regionaux de pharmacovigilance. [Psychiatric disorders associated with montelukast: data from the National Pharmacovigilance Database]. Arch Pediatr. 2013 Mar;20(3):269-73. doi: 10.1016/j.arcped.2012.12.006. Epub 2013 Feb 1. French. PMID 23375423